CLINICAL TRIAL: NCT01329809
Title: A Phase IIa Study of Neoadjuvant JX-594 (Thymidine Kinase-Deactivated Vaccinia Virus Plus GM-CSF) Administered by Intravenous Infusion or Intratumoral Injection Followed by Surgical Resection in Patients With Metastatic Colorectal Tumors Within the Liver
Brief Title: Neoadjuvant Study of Recombinant Vaccinia Virus to Treat Metastatic Colorectal Carcinoma in Patients Undergoing Complete Resection of Liver Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Jennerex Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JX594-HEP012
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2011-07

CONDITIONS: Colorectal Carcinoma
Keywords: metastatic colorectal cancer; colon cancer; liver metastasis; Pexa-vec; JX-594
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JX-594 Intravenous infusion (Experimental): JX-594 will be administered intravenously to patients with measurable intra-hepatic disease who are not eligible for intratumoral injection of JX-594.
  Interventions: Drug: Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594)
- JX-594 Intratumoral Injection (Experimental): JX-594 will be injected directly into the liver tumor of patients who have at least two measurable intra-hepatic tumors, one of which must be at least 1.5cm in diameter and safety injectable.
  Interventions: Drug: Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594)

INTERVENTIONS:
Drug: Recombinant Vaccinia GM-CSF; RAC VAC GM-CSF (JX-594) — intratumoral or intravenous dosage: 10e9 pfu Intravenous: administered over 60 minutes Intratumoral: direct injection into a single liver lesion
  Other Names: JX-594

SUMMARY:
This is a neoadjuvant Phase 2a, open-label trial in patients with metastatic colorectal carcinoma who are undergoing a complete resection of the metastatic colorectal tumors in their liver.

DETAILED DESCRIPTION:
Patients will receive either an intravenous infusion or an intratumoral injection of JX-594 (Pexa-Vec) directly into one liver lesions at Day 1. Patients will undergo a complete resection of all liver tumors at Day 15. Patients will then be monitored throughout their life for disease recurrence and/or general overall survival.

ELIGIBILITY:
Inclusion Criteria:

* The planned surgical resection must be margin negative with complete resection or resection plus radiofrequency ablation (RFA) of metastatic CRC as determined by principal investigator or surgeon
* Diagnosis of histologically-confirmed metastatic colorectal tumor(s) within the liver eligible for surgical resection. Eligible patients must have: preoperative work-up that reveals potential resectability (CT scan or MRI of the abdomen and pelvis and CT scan of the chest within 6 weeks of enrollment) preoperative work-up to ensure operability with general medical clearance as indicated
* At least one measurable tumor mass by MRI (i.e. lesion that can accurately be measured in at least one dimension with longest diameter ≥ 1 cm)
* Plan for a maximum resection of six (6) liver segments
* Child Pugh A (Refer to APPENDIX C: Child-Pugh Classification
* Performance Score: KPS score of ≥ 70
* Age ≥18 years
* For patients treated with IT injection only: at least 1 intra-hepatic tumor with longest diameter (LD) ≥ 1.5 cm and ≤ 12 cm and which is technically amenable to injection under radiographic guidance targeted for surgical resection.
* In patients treated with IT injection, the injected tumor must be included in the surgical resection specimen (a planned RFA of the injected tumor would not be eligible)
* Total bilirubin ≤ 3 x ULN
* AST, ALT < 5.0 x ULN
* WBC ≥ 3.5x 109/L and ≤ 50 x 109/L
* ANC ≥1.5 x 109/L
* CD4 ≥ 200 total cells/mm3
* Hemoglobin ≥ 80g/L
* Platelet count ≥ 100 x 109/L
* Acceptable coagulation status: INR ≤ 1.4
* Creatinine ≤ 2 x ULN
* Serum Sodium, Potassium and Calcium levels ≤ Grade 1
* If patients are diabetic or have a screening random glucose > 8.9mmol/L, a fasting glucose must be done and results must be WNL or Grade 1 in order to be eligible for the study.
* For patients who are sexually active: patient must be able and willing to abstain from sex during JX-594 treatment period (to prevent pregnancy) and willing to use barrier method for at least 6 weeks after the last JX-594 treatment (to protect partner against infection).
* Able and willing to sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)/Research Ethics Board (REB)-approved written consent form Able and willing to comply with study procedures and follow-up examinations, including compliance with the "Infection Control Guidelines for Patients" contained within the written consent form.

Exclusion Criteria:

* Prior local-regional treatment (including hepatic arterial infusion, hepatic embolization, radiofrequency ablation) for tumor downstaging. Prior adjuvant chemotherapy will be accepted as long as the duration between chemotherapy and the development of metastases has been >8 weeks.
* Pregnant or nursing an infant
* Known myeloproliferative disorders requiring systemic therapy
* Significant immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or medication (e.g. high dose systemic corticosteroids taken for more than 4 weeks within the preceding 3 months)
* History of severe exfoliative skin condition (e.g. eczema or atopic dermatitis requiring systemic therapy for more than 4 weeks)
* Tumor(s) invading a major vascular structure (e.g. carotid artery)
* Clinically significant and/or rapidly accumulating ascites, pericardial and/or pleural effusions
* Clinically significant active infection, requiring systemic antibiotic therapy, or uncontrolled medical condition which would, in the opinion of the principle investigator, impair the ability of the subject to receive protocol therapy
* Severe or unstable cardiac disease, including significant coronary artery disease requiring angioplasty or stenting within the preceding 12 months, unless well-controlled and on stable medical therapy for at least 3 months
* Known viable CNS malignancy (history of completely resected or irradiated brain metastases allowed)
* Chronic use of anti-platelet or anti-coagulation medication that cannot be temporarily discontinued for at least seven days prior to treatment with JX-594. (Note: the following are allowed: low dose aspirin ≤ 100 mg, low dose coumadin as long as INR ≤ 1.4 and low-dose heparin to maintain port access)
* Use of the following anti-viral agents: ribavirin, adefovir, cidofovir (at least 7 days prior to the first treatment), and PEG-IFN (at least 14 days prior to the first treatment).
* Absolute contraindication to undergoing MRI scanning (e.g. pacemaker, paramagnetic intracranial aneurysm clip, inner ear implants, fragments of metal within the body, etc.).
* Pulse oximetry O2 saturation < 90% at rest
* Experienced a severe systemic reaction or side-effect as a result of a previous smallpox vaccination
* Inability or unwillingness to give informed consent or comply with the procedures required in this protocol.
* Patients with household contacts who meet any of these criteria will be excluded unless alternate living arrangements can be made during the patient's dosing period and for at least 7 days following the last dose of study medication
* Pregnant or nursing an infant
* Children < 1 year old
* People with skin disease (eczema, atopic dermatitis and related diseases
* Immunocompromised hosts (severe deficiencies in cell-mediated immunity, including AIDS, organ transplant recipients, hematologist malignancies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Delivery to and replication within tumors | Day 1, 3, 5, 8, 11, and 15
  IT injection: replication and dissemination of JX-594 following injection of a single colorectal metastasis within the liver. A positive replication response is defined as a > 2-fold increase in viral genome concentration in the blood(as measured in the first 12 hours following injection) within the first 14 days following treatment.
  Note: Viral genomes will be measured in the blood by Q-PCR at baseline, on Day 1 (15 minutes, 3 hours & 8 hours) post-treatment and on Days 3, 5, 8, 11 and 15.
  IV infusion: assessment of viral gene & protein expression in histologic samples of tumor tissue

SECONDARY OUTCOMES:
JX-594 spread to, and replication within, non-injected tumors after IT JX-594 injection | Day 1
  JX-594 spread to, and replication within, non-injected tumors after IT JX-594 injection as measured by the presence of viral protein expression and/or LacZ expression in non-injected tumor sections from at least 1) two different non-consecutive cuts, both of which contain viable tumor tissue in at least 10 high power fields; and 2) at least 5 cells in one high power field show positive staining for viral protein and/ or LacZ expression
Modified Choi response assessment | Day 8-14
  Modified Choi response assessment based on DCE-MRI at baseline and between Days 8 14 (within 7 days prior to surgical resection)
Toxicity: Grade I-IV Adverse Events (according to CTCAE) | Day 1- Day 43
  Toxicity: Grade I-IV Adverse Events (according to CTCAE); including surgical complications such as delay of surgery, prolonged hospitalization, bleeding (monitor transfusion requirements), postoperative infections, bile leak, hepatic failure sepsis and death

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Auer, MD, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital and Research Institute (OHRI), Ottawa, Ontario, Canada